CLINICAL TRIAL: NCT06743425
Title: A Pilot Study of a Remote Attention-Deficit/Hyperactivity Disorder Monitoring Program (RAMP) for Children in Rural Areas
Brief Title: A Pilot Study of a Remote ADHD Monitoring Program
Acronym: RAMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IDeA States Pediatric Clinical Trials Network (Network)
Collaborators: Medical University of South Carolina (Other); University of Mississippi Medical Center (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 276280
Record Dates: First submitted 2024-12-11; First posted 2024-12-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Attention-deficit/Hyperactivity Disorder; ADHD
Keywords: Rural health; Vanderbilt; Text-based Symptom Reporting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a multi-center, parallel, unblinded, randomized controlled clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAMP Reports (Experimental): Submit RAMP reports weekly for 4 weeks and then monthly for 2 months.
  Interventions: Other: RAMP Reports
- Digital Education Handouts (Active Comparator): Standard of care determined by the treating healthcare provider and digital education handouts (attention controls) distributed by the study team weekly for 4 weeks and then monthly for 2 months.
  Interventions: Other: Digital Education Handouts

INTERVENTIONS:
Other: RAMP Reports — Participants will receive text-based requests for reports with embedded links to select radio button questionnaires directly on their mobile device. Questions include current inattention/hyperactivity symptoms, school performance, and any engagement in behavioral therapy. Inattention/hyperactivity symptom questions and scoring is taken directly from the publicly available Vanderbilt Rating Scales, which is a commonly used, guideline-recommended tool for both diagnosis and management of ADHD for use by parents and teachers.
  Other Names: Remote ADHD Monitoring Program
  Arms: RAMP Reports
Other: Digital Education Handouts — The digital education handouts will be sent via email to the control group and will serve as an attention control. They will consist of information regarding a general pediatric health topic and will be emailed at intervals matching the RAMP requests in the intervention group.
  Other Names: Standard of Care
  Arms: Digital Education Handouts

SUMMARY:
RAMP is a pilot study examining the use of an Attention-Deficit/Hyperactivity Disorder (ADHD) Monitoring Program during the early stages of treating ADHD in children living in rural settings. This trial will enroll 36 caregiver/infant dyads across 2 sites and will evaluate feasibility endpoints rather than clinical outcomes. Enrolled participants will be randomized 1:1 to the intervention group (RAMP reports) or control group (digital education handouts). The study duration is 10 months, including start-up, enrollment and intervention, and data analysis and manuscript submission.

DETAILED DESCRIPTION:
The RAMP study is designed to examine the use of an attention-Deficit/Hyperactivity Disorder (ADHD) Monitoring Program during the early stages of treating ADHD in children living in rural settings. It is a multi-site pilot study conducted across two Institutional Development Award (IDeA) States Pediatric Clinical Trials Network (ISPCTN) sites in conjunction with four practices with high rural and/or underserved populations.

The Remote ADHD Monitoring Program (RAMP) will include provider ADHD Best Practice education, caregiver and teacher prompts for frequent RAMP Reports of inattention and hyperactivity symptoms and a provider dashboard with enrolled children. The RAMP Report includes the publicly available Vanderbilt Rating Scales (henceforth shortened to Vanderbilt Assessment), which is a commonly used, guideline-recommended tool for both diagnosis and management of ADHD for use by parents and teachers.

Families will be approached until 36 caregiver/child dyads are enrolled. Those enrolled will be randomized 1:1 to either the intervention group or control group. The intervention group will be enrolled in the RAMP, with prompts to provide frequent reports including ADHD symptoms. The control group will provide ADHD symptom reports through paper forms (usual care), on a provider determined schedule.

The intervention group will be enrolled in the RAMP platform and will receive text-based requests for reports with embedded links to fill out the RAMP questionnaires weekly for 4 weeks, then monthly for 2 months. The control group will receive digital education handouts about age-appropriate pediatric health topics weekly for 4 weeks, then monthly for 2 months.

For the intervention group, the child's teacher can voluntarily return the RAMP questionnaires as well, but will not have direct contact with the study team. The child's provider will also be a participant for the intervention group, and will receive requests to review the submitted RAMP reports.

The primary endpoint for this study is to evaluate the number of clinical assessments per participant that are completed by caregivers and teacher and returned to providers for ADHD management.

The secondary endpoint for this study is to evaluate the proportion of all submitted RAMP reports that are reviewed by providers.

The results of this pilot will be used to design a full-scale efficacy trial in additional rural sites to expand diversity and assess generalizability.

ELIGIBILITY:
Inclusion Criteria:

The child must

* be under the care of a participating provider
* be aged 5-11 at enrollment
* have a diagnosis of ADHD
* be initiating stimulant medication for treatment for the first time or have not received stimulant medication for the last 6 months
* be attending in-person elementary school

The Primary caregiver must

* be willing and legally able to give consent
* have access to a smartphone
* be English-speaking
* reside with the child at least 3 days per week
* complete an initial symptom assessment prior to starting stimulant treatment and be willing to provide a copy to the study team

The provider must

* manage ADHD care in patients age 5-11 years
* provide informed consent
* agree to use the RAMP platform if they care for patients randomized to use it
* agree to provide information to potential participants about the study and contact the research coordinator if interested

Exclusion Criteria:

Child:

* has serious mental health comorbidities (Children with depression, anxiety, oppositional defiant disorder will be permitted to participate. Children with schizophrenia, bipolar disorder, conduct disorder and those who have been hospitalized for any mental health condition will be excluded from the study.)
* has severe neurodevelopment disorders (Children with well-controlled seizure disorders will be permitted to participate.)
* is currently receiving, or previously received, atypical antipsychotic medication treatment
* is or becomes pregnant

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate completion of clinical assessments by caregivers and teachers. | 6 Months
  The number of clinical assessments (paper assessments in control and RAMP Reports in intervention) per participant that are completed by caregivers and teachers and returned to providers for ADHD management.

SECONDARY OUTCOMES:
Evaluate provider acceptability of the RAMP through utilization measures. | 6 Months
  The proportion of all submitted RAMP Reports that are reviewed by providers.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Investigators will conduct this trial following the publication and data-sharing policies and regulations listed below:
  NIH Public Access Policy requires scientists to submit final peer-reviewed journal manuscripts arising from NIH funds to the digital archive PubMed Central upon acceptance for publication.
  Environmental Influences on Child Health Outcomes (ECHO) IDeA States Pediatric Clinical Trials Network (ISPCTN) Publications and Presentations Policy ensures the accurate, responsible, and efficient communication of findings from ECHO ISPCTN clinical trials.
  NIH Data Sharing Policy and the policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Resulting Information Submission Rule. Other researchers may request data from this trial by contacting Song Ounpraseuth, Ph.D., at the ISPCTN Data Coordinating and Operations Center (DCOC).
Supporting Information: SAP, ICF
Time Frame: Per data sharing polices of NIH and the ISPCTN

REFERENCES:
- [Derived] MacGeorge CA, Henry M, Ford HA, Malloch L, Fratesi E, Cabaniss S, Baldner J, Greer M, Gaffney K, Bimali M, Abraham P, Fu LY, Ounpraseuth PS, Turley CB. Study protocol for a pilot study for Remote ADHD Monitoring Program (RAMP) for children in rural areas. PLoS One. 2025 Dec 2;20(12):e0337802. doi: 10.1371/journal.pone.0337802. eCollection 2025. PMID 41329787